CLINICAL TRIAL: NCT03220360
Title: Application of Different Biomaterials in the Preservation of Vital Pulp in Carious Deciduous Teeth: a Prospective, Single-center, Randomized, Controlled Clinical Trial
Brief Title: Application of Different Biomaterials in the Preservation of Vital Pulp in Carious Deciduous Teeth
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Chengdu Maternal and Children's Health Care Hospital (Other)
Responsible Party: Principal Investigator, Xiaohong Ma, Principal Investigator, Chengdu Maternal and Children's Health Care Hospital
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Treatment
Other Study IDs: ChengduMCHCH-001
Record Dates: First submitted 2017-07-14; First posted 2017-07-18 (Actual); Last update posted 2017-07-18 (Actual); Status verified 2017-07

CONDITIONS: Tooth, Deciduous

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- indirect pulp capping group (Experimental): Sixty children with deep caries of deciduous teeth underwent indirect pulp capping, and they were selected and randomized into four groups according to pulp capping agents: MTA group, calcium hydroxide group, Biodentine group and TheraCal group.
  Interventions: Procedure: indirect pulp capping
- direct pulp capping group (Experimental): Sixty children with deep caries of deciduous teeth underwent direct pulp capping, and they were selected and randomized into four groups according to pulp capping agents: MTA group, calcium hydroxide group, Biodentine group and TheraCal group.
  Interventions: Procedure: direct pulp capping
- vital pulpotomy group (Experimental): Forty-five children with deep caries of deciduous teeth underwent vital pulpotomy, and they were selected and randomized into four groups according to pulp capping agents: MTA group, calcium hydroxide group, Biodentine group and TheraCal group.
  Interventions: Procedure: vital pulpotomy

INTERVENTIONS:
Procedure: indirect pulp capping — Sixty children with deep caries of deciduous teeth underwent indirect pulp capping and they were selected and randomized into four groups according to pulp capping agents: MTA group, calcium hydroxide group, Biodentine group and TheraCal group.
  Arms: indirect pulp capping group
Procedure: direct pulp capping — Sixty children with deep caries of deciduous teeth underwent direct pulp capping and they were selected and randomized into four groups according to pulp capping agents: MTA group, calcium hydroxide group, Biodentine group and TheraCal group.
  Arms: direct pulp capping group
Procedure: vital pulpotomy — Forty-five children with deep caries of deciduous teeth underwent vital pulpotomy and they were selected and randomized into four groups according to pulp capping agents: MTA group, calcium hydroxide group, Biodentine group and TheraCal group.
  Arms: vital pulpotomy group

SUMMARY:
To compare the efficacies of MTA, calcium hydroxide preparation, Biodentine and TheraCal LC that are commonly used in pediatric dentistry in the preservation of vital pulp in carious deciduous teeth.

DETAILED DESCRIPTION:
In recent years, the importance of deciduous teeth and the hazards of caries in deciduous teeth have gradually attracted the attention of professionals and parents of children. The dental pulp disease and periapical disease of deciduous teeth are the main and important factors that cause deciduous teeth defects, deciduous dentition and mixed dentition deletion, which have a serious impact on the physical and mental health of children from the local or systemic aspects. From the point of view of children's stomatology, according to the principle of treatment of dental caries of deciduous teeth, vital pulp preservation should be selected in patients with deep caries and reversible pulpitis; This concept has been carried forward especially after the advent of new materials with good biocompatibility and good edge sealing. After judging the existing state of the affected teeth (such as deep caries or reversible pulpitis) and removal of caries, indirect pulp capping, direct pulp capping, and vital pulpotomy can be correspondingly selected. Complete healthy pulp can be preserved in indirect pulp capping and direct pulp capping. During vital pulpotomy, coronal pulp due to infection induced by various causes is removed, and healthy root pulp is retained.

The success of the preservation of vital pulp in carious deciduous teeth depends not only on determining the health status of the pulp, but also on selecting the most suitable pulp capping agent. No matter the use of calcium hydroxide and mineral trioxide aggregate (MTA) or new biomaterials, controlling pulp inflammation and preserving healthy pulp are the keys to successful treatment. The clinical reality is that it is not easy to determine the state of the pulp accurately because of the child's feelings of pain and the unreliability of the description. Thus, the secondary treatment can be easily produced after treatment. For example, pulp re-infection requires dental pulp extraction; or severe infection results in removal of the affected teeth and space maintenance. In the face of this reality, many clinicians will advise parents to select dental pulp extraction for deciduous teeth at the first visit. If there is a reliable clinical pathway for the preservation of the vital pulp of the carious deciduous teeth, the doctor will put aside his worries. Therefore, this study is designed to find a suitable clinical pathway and to increase the success rate of the preservation of the vital pulp of carious deciduous teeth. The key to solving this problem lies in the selection of suitable pulp capping agent, as well as the repair method of the crown selection to obtain a better edge sealing. Numerous studies have confirmed that crown repair of deciduous teeth can obtain better edge sealing on the basis of obtaining the largest degree of morphological restoration. The difficulty and key point are to select the best biomaterials as the pulp capping agents for the preservation of vital pulp.

The investigators will select classical and new biomaterials for the preservation of vital pulp and compare them so as to select a pulp capping agent with high success rate. With the further research of biomedical ceramic materials, such as restorative material for pulposis Bioaggregate and restorative material to dentin Biodentine, the biocompatibility of such materials allows the destructed dental pulp tissue to be reconstructed. Shayegan et al. performed vital pulpotomy for pigs using Biodentine, white MTA and formaldehyde cresol as pulp capping agents, and using Biodentine, white MTA and calcium hydroxide as direct pulp capping, and observed the response to dental pulp tissue. They concluded that Biodentine and white MTA have the same biocompatibility, and they are suitable for the pulp capping material of porcine deciduous teeth. In recent years, TheraCal LC has emerged as a new type of pulp capping agent. Some scholars believed that both MTA and TheraCal are good indirect pulp capping materials. TheraCal has better operability and similar chemical property as MTA. In the indirect pulp capping treatment of deciduous teeth, TheraCal can be a successful alternative to MTA. Nevertheless, TheraCal is rarely used in direct pulp capping, and vital pulpotomy.

In summary, this study will select Biodentine and TheraCal, verify their efficacies, and explore their superiorities. Calcium hydroxide and MTA will be selected as controls, which will be separately used in indirect pulp capping, direct pulp capping, and vital pulpotomy to provide reliable choices for clinicians.

ELIGIBILITY:
Inclusion Criteria:

* Indirect pulp capping or direct pulp capping: (1) Patients from Chengdu Maternal and Child Center, China; (2) Age between 4 and 7 years old; (3) The affected teeth present healthy periodontal occlusion or adjacent deep caries; (4) no history of spontaneous pain, root length more than 2/3, without periapical lesions and sinus; (5) written informed consent is provided by parents or guardian after they indicate that they fully understand the treatment plan.
* Vital pulpotomy: (1) Patients from Chengdu Maternal and Child Center, China; (2) Age between 3 and 8 years old; (3) mandibular deciduous molars with deep caries; (4) all the affected teeth are in the stable phase of tooth root; (5) written informed consent is provided by parents or guardian after they indicate that they fully understand the treatment plan.
* Blank control teeth: (1) The normal teeth on the opposite side of the teeth will be chosen as blank controls; (2) no dental caries; (3) X-ray films reveal that bifurcation and periapical area do not present shadow, and tooth root is also in stable period; (4) written informed consent is provided by parents or guardian after they indicate that they fully understand the treatment plan.

Exclusion Criteria:

* Patients with one or more of the following conditions will be excluded from this study.
* Dental pulp lesions, tooth resorption, pulp calcification, root tip or root furcation.

Ages: 3 Years to 8 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 165 (Actual)
Dates: Start 2016-06-01 (Actual); Primary Completion 2017-09 (Estimated); Study Completion 2018-09 (Estimated)

PRIMARY OUTCOMES:
image findings | at month 12 after surgery
  To observe thickness of reparative dentin. Image data are processed by XCP technology, scanned and transferred to a computer for digital analysis, preoperative reference value is used as the basis.

SECONDARY OUTCOMES:
degree of root resorption | at month 12 after surgery
  Degree of root resorption: ①Zero: no abnormal root resorption; ②mild: root resorption accounts for less than 1/4 of root length; ③moderate: root resorption accounts for 1/4-1/2 of root length; ④severe: root resorption accounts for more than 1/2 of root length.

IPD SHARING:
Plan to Share IPD: Undecided